CLINICAL TRIAL: NCT01622309
Title: Effect of Balanced Hypocaloric Diet Associated With Supplementation of Eggplant Meal in the Remission of Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Mauara Scorsatto, Doctoral student, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 062/10-CEP
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Obesity, Abdominal
Keywords: Oxidative Stress; Obesity; Solanum melongena
MeSH Terms: conditions — Obesity; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- eggplant meal (Active Comparator): 13 g meal of eggplant/day
  Interventions: Dietary Supplement: eggplant meal
- cassava meal (Placebo Comparator): 13 g of placebo/day
  Interventions: Other: cassava meal

INTERVENTIONS:
Dietary Supplement: eggplant meal — 13 g meal of eggplant/day, being 6,5 g in breakfast and 6,5g in dinner
  Arms: eggplant meal
Other: cassava meal — 13g cassava meal/day,being 6,5 g in breakfast and 6,5g in dinner
  Arms: cassava meal

SUMMARY:
Cardiovascular diseases (CVD) prevail as the main cause of death in developed and developing countries and are among the most frequent causes of disabilities in Brazil and in the world.

Economic alternatives have been studied to assist in reducing cardiovascular risk factors. Within this context, the Solanum menogena, whose fruit known as eggplant is widely consumed in Brazil, is being used in alternative medicine with the purpose to reduce the concentrations of cholesterol, glucose and promote loss of body weight.

Aubergine (eggplant) stands out for its high fibre content (approximately 40%) and low fat content. In addition, it is popularly known for its functional properties, aiding in reducing the risk of coronary diseases. The purplish coloring of the eggplant peel is attributed to the large amount of flavonoids, which have antioxidant properties and contribute to the flavor of eggplant.

The investigators hypothesis is that the eggplant flour associated with a restricted calorie diet has effect in reduction in waist circumference, reduction of body fat and increasing HDL-cholesterol; this way, contributing to the reduction of cardiovascular risk factors

All participants will be informed about the research and they will have to sign a consent form. The volunteers will be divided into two groups: one group will receive a restricted-calorie diet and supplementation with eggplant flour; and the other will receive a diet plus a placebo for 120 days, being both groups evaluated monthly. In each consultation, evaluation of weight, body composition, fulfillment of the diet and blood pressure measurement will be performed. In addition, blood will also be collected in order to determine glucose, insulin, total cholesterol, LDL, HDL, triglycerides, oxidized anti-LDL antibodies, 15-isoprostane and minerals (selenium, zinc, iron, manganese, magnesium and copper). The results will be analyzed by statistical program.

The investigators expect that with the results obtained, the eggplant flour can be used as an ally in the prevention of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

adults (aged> 20 years) body mass index (BMI)> 25 kg/m2 for both sexes, of any ethnicity.

Exclusion Criteria:

smokers, pregnant women, nursing mothers and that are performing diets and / or using drugs for weight reduction and supplements of any kind.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Increasing cholesterol- HDL of 10% | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Policlínica de Alcantara, São Gonçalo, Rio de Janeiro, Brazil